CLINICAL TRIAL: NCT03066765
Title: Non-Randomized, Single Arm Study of the New Linguaflex Tongue Retractor for the Treatment of Obstructive Sleep Apnea
Brief Title: LTR for Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linguaflex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTR-005-V01.2
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LTR Treatment (Experimental): An implant device (Linguaflex Tongue Retractor) will be placed in the tongue and assessed for safety and efficacy
  Interventions: Device: Linguaflex Tongue Retractor

INTERVENTIONS:
Device: Linguaflex Tongue Retractor — Tongue implant

SUMMARY:
Study of tongue implant for treatment of obstructive sleep apnea

DETAILED DESCRIPTION:
Subjects with obstructive sleep apnea will be treated with a tongue based suspension implant technique to keep airway open while sleeping. Subjects will be followed a year with primary endpoint of AHI results through Polysomnography readings (PSG) testing in an overnight sleep lab.

ELIGIBILITY:
Inclusion Criteria:

* AHI>10
* 18 years of age

Exclusion Criteria:

* Subjects with >20% of their AHI accounted for from central apnea.
* Mallampanti score of 4
* Tonsillar hypertrophy (4+)
* Prior uvulopalatopharyngoplasty (UPPP) procedure
* Narrowing of hypopharynx airspace more than velopharyngeal airspace as seen on examination or x-ray
* Tongue thickness <40 mm measured on lateral cephalogram x-ray from the frenulum to linea terminalis
* More than 10% of sleep time with blood O2 desaturation below 70%
* Unable and/or unwilling to comply with study requirements
* Females of child bearing age who are pregnant or intending to become pregnant
* Allergy to silicone
* History of radiation therapy to neck or upper respiratory tract
* Subjects with bleeding disorders, impaired immunity for any reason, or heart attack within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with AHI decrease greater than or equal to 50% and less than a score of 10 according to PSG testing | 1 year
  Recording of Apnea Hypopnea Index through polysomnography during overnight sleep study

SECONDARY OUTCOMES:
Number of subjects of Adverse Events and Serious Adverse Events through recording number, type and relation to device | 1 year
  Assessment of Adverse Events and Serious Adverse Events
Number of subjects with significant change in sleepiness and score of less than 10 using Epworth Sleep Scale | 1 year
  Assess level of sleepiness pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Balwinder Singh, MD, Principal Investigator — Putrajaya Hospital

IPD SHARING:
Plan to Share IPD: No